CLINICAL TRIAL: NCT00057616
Title: Multicenter, Randomized, Double-blind, Placebo-controlled Study to Compare the Efficacy and Safety of CC-5013 vs. Placebo in Subjects With Metastatic Malignant Melanoma Whose Disease Has Progressed on Treatment With DTIC, IL-2, or IFN Based Therapy
Brief Title: Study to Compare the Efficacy and Safety of CC-5013 vs. Placebo in Subjects With Metastatic Malignant Melanoma.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CC-5013-MEL-002; NCT00051064 (obsolete NCT alias)
Record Dates: First submitted 2003-04-04; First posted 2003-04-07 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Melanoma; Neoplasm Metastasis
Keywords: Metastatic Melanoma; Melanoma; Revimid; CC5013
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — Lenalidomide

INTERVENTIONS:
Drug: CC-5013

SUMMARY:
Subjects are randomized to one of two treatment arms. All subjects are screened for eligibility within 28 days prior to randomization. The study consists of a treatment phase and a follow-up phase. Subjects are treated in repeating 4 week cycles.

ELIGIBILITY:
* Understand and voluntarily sign an informed consent form
* Able to adhere to the study visit schedule and other protocol requirements
* Metastatic malignant melanoma now stage IV, relapsed or refractory to standard metastatic therapy
* Women of childbearing potential must have a negative serum or urine pregnancy test within 7 days of starting study drug
* Patients with active brain disease, or newly diagnosed brain metastases, within 4 weeks prior to the start of study treatment are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274
Dates: Start 2002-10-01 (Actual); Study Completion 2005-07-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (49):
- Australia (12):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Sydney Cancer Centre, Camperdown, New South Wales
  - Royal Newcastle Hospital, Newcastle, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Roayl Brisbane Hospital, Herston, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Cabrini Hospital, Malvern, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Mount HospitalOncology, Perth, Western Australia
- Estonia (2):
  - North-Estonian Regional Hospital, Tallinn
  - Tartu University Clinics Onkology & Haematology Clinic, Tartu
- Germany (7):
  - Klinick fur Dermatologie, Berlin
  - Dermatologie Klinik der Ruhr Universitat Bochum- St. Joseph's Hospital, Bochum
  - Klinick fur Dermatolgie, Bonn
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - Universitatsklinik Eppendorf, Hamburg
  - Kinkum der Christian-Albrecht-Universitat KielDepartment of Dermatologie, Kiel
  - Klinik fur DermatologieVenerologie und Allergologie, Mannheim
- Latvian Onkology Centre, Riga, Latvia
- Lithuania (2):
  - Klaipeda Hospital, Klaipėda
  - Vilnius University Onkology Institute, Vilnius
- Daniel DenHoed Kliniek, Rotterdam, Netherlands
- South Africa (8):
  - Panorama Medi-Clinic / Panorama Oncology Unit, Cape Town
  - Addington Hospital, Durban
  - Wilgers Hospital / Wilgers Oncology Centre, Hatfield, Pretoria
  - Sandton Oncology Centre, Morningside, Johannesburg
  - St. Georges Hospital, Port Elizabeth
  - Little Company of Mary / Mary Potter Oncology Centre, Pretoria
  - Pretoria Academic Hospital / Department Medical Oncology, Pretoria
  - Durban Oncology Centre, Westridge, Durban
- Ukraine (7):
  - Dnipropetrovsk State Medical Academy, Dnipropetrovsk
  - Kharkov Postgraduate Medical Academy, Kharkov Regional Clinical Oncology Center, Kharkiv
  - Scientific Research Institute of OncologySoft Tissue Department, Kiev
  - Kiev City Oncology Hospital, Kiev
  - Lviv State Medical University Regional Oncology Centre, Lviv
  - Odessa Regional Oncology DispensaryChemotherapy Dept, Odesa
  - Uzhgorod Regional Oncology Diepensary, Uzhhorod
- United Kingdom (9):
  - Cancer Centre, Egbaston, Birmingham
  - Christies Hospital, Withington, Manchester
  - Beatson Oncology CentreWestern InfirmaryOncology, Glasgow
  - Cancer Research BldgDivsion of Cancer Medicine Research, Leeds
  - Roayl Free Hospital, London
  - St. George's Hospital, London
  - Royal Marsden Hospital Department of Oncology, London
  - Royal Marsden Hospital, London
  - Newcastle GeneralOncology, Newcastle

REFERENCES:
- [Background] Eisen T, Trefzer U, Hamilton A, Hersey P, Millward M, Knight RD, Jungnelius JU, Glaspy J. Results of a multicenter, randomized, double-blind phase 2/3 study of lenalidomide in the treatment of pretreated relapsed or refractory metastatic malignant melanoma. Cancer. 2010 Jan 1;116(1):146-54. doi: 10.1002/cncr.24686. PMID 19862820